CLINICAL TRIAL: NCT00992251
Title: A Prospective, Single Product, Observational Registry Involving Patients Presenting With Locally Advanced or Metastatic Prostate Cancer Receiving Eligard as Androgen Deprivation Treatment.
Brief Title: Eligard Observational Registry for Patients With Prostate Cancer
Status: Completed | Type: Observational
Sponsor: CMX Research (Other)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor
Other Study IDs: LEUPR_L_04620
Record Dates: First submitted 2009-10-07; First posted 2009-10-09 (Estimated); Last update posted 2016-12-22 (Estimated); Status verified 2016-12

CONDITIONS: Cancer of the Prostate
Keywords: prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The objective of this registry is to collect data on patient demographics, medical history, change in prostate, bone and overall health of the patients receiving androgen ablation treatment using Eligard. Data collected through this national registry program provides an opportunity to increase knowledge of efficacy and safety of the long term treatment with Eligard, provide a platform to better identify patient segments for the therapy with Eligard®. Furthermore registries are the only tools to accurately capture rare adverse events.

DETAILED DESCRIPTION:
354 patients were enrolled in this study. Only 88 patients completed the study.

For those patients completing the three years of data collection, 10% were considered Castrate Resistant and remained on Eligard®. For those patients not completing 3 years of follow-up, 8.8% were considered Castrate Resistant and did not continue in the study.

ELIGIBILITY:
Inclusion Criteria:

* Patients > 18 years of age.
* Histologically confirmed diagnosis of locally Advanced or Metastatic Prostate Cancer.
* Patient starting an androgen deprivation therapy with Eligard at 3 or 4 month treatment frequency per standard of care.
* Signed written informed consent.

Exclusion Criteria:

* Prior ADT (within 6 months).
* Any concurrent condition that would make it undesirable, in the physician's opinion, for the subject to participate in the study or would jeopardize compliance with the protocol.
* Life expectancy less than 2 years.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients > 18 years of age. Histologically confirmed diagnosis of locally Advanced or Metastatic Prostate Cancer Patient starting an androgen deprivation therapy with Eligard at 3 or 4 month treatment frequency per standard of care.
Sampling Method: Non-Probability Sample
Enrollment: 354 (Actual)
Dates: Start 2009-08; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Determine the percentage of patients that will achieve a hormone refractory status at 3 years after initiation of Androgen Deprivation Treatment with Eligard®. | 3 Years

SECONDARY OUTCOMES:
Determine what baseline patient characteristics are associated with becoming hormone refractory at 3 years. | 3 years
Collect data on patient demographics, medical history, and change in prostate-, bone- and overall health of the patients receiving androgen ablation treatment using Eligard®. | 3 years
Collect referral data if the patient was referred to a medical oncologist during treatment. | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Hélène Grassin, Study Director — Sanofi
Locations (36):
- Canada (36):
  - Dr. George Vrabec, Abbotsford, British Columbia
  - Southern Interior Medical Research Corporation, Kelowna, British Columbia
  - Dr. Cal Andreou, Surrey, British Columbia
  - Dr. Nazif Omar, Surrey, British Columbia
  - Dr. Herman Kwan, Surrey, British Columbia
  - Dr. Joseph Zadra, Barrie, Ontario
  - Dr. Jonathan Giddens, Brampton, Ontario
  - Brantford Urology Research, Medical Arts Building, Brantford, Ontario
  - G. Kenneth Jansz Medicine Professional Corporation, Burlington, Ontario
  - Dr. Bisshwajit Bora, Greater Sudbury, Ontario
  - Dr. Eric Hirshberg, Guelph, Ontario
  - Dr. Anil Dapoor, Hamilton, Ontario
  - Dr. Giovanni A. DiCostanzo, Markham, Ontario
  - Dr. Morrie Liquornik, Newmarket, Ontario
  - Dr. Roger Buckley, North York, Ontario
  - Dr. Stanley Flax, North York, Ontario
  - Dr. Jack Barkin, North York, Ontario
  - Dr. Richard Casey, Oakville, Ontario
  - Orillia Urology Associates, Orillia, Ontario
  - Kawartha Urology Associates, Peterborough, Ontario
  - Dr. Mohamed Elharram, Peterborough, Ontario
  - Dr. Emmanuel Abara, Richmond Hill, Ontario
  - Dr. Vinod Mathur, Sault Ste. Marie, Ontario
  - Dr. Edward Woods, Scarborough Village, Ontario
  - Dr. Nick Logarakis, Toronto, Ontario
  - Dr. Harold Kwok, Toronto, Ontario
  - Dr. Ashis Chawla, Toronto, Ontario
  - Dr. Jain Umesh, Toronto, Ontario
  - Dr. Louis-Rene Barrette, Chicoutimi, Quebec
  - Dr. Mahmoud Nachabe, Greenfield Park, Quebec
  - Polyclinique Med Concorde, Laval, Quebec
  - Dr. Thu Van Nguyen, Montreal, Quebec
  - Dr. Pierre Karakiewicz, Montreal, Quebec
  - Dr. John Vary, Rimouski, Quebec
  - Dr. Thierry Tremblay, Val-d'Or, Quebec
  - Westmount Med Bldg, Westmount, Quebec

IPD SHARING:
Plan to Share IPD: Undecided